CLINICAL TRIAL: NCT01386112
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Safety and Tolerability Phase 1/2a Study of Two Dosing Regimens of EUR-1100 for Oral Use, in Subjects With Eosinophilic Esophagitis (EoE)
Brief Title: Safety and Tolerability Study of Oral EUR-1100 to Treat Eosinophilic Esophagitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-021
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- EUR-1100 1.5 mg (Experimental)
  Interventions: Drug: EUR-1100
- EUR-1100 3.0 mg (Experimental)
  Interventions: Drug: EUR-1100
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: EUR-1100 — Active oral medication
  Arms: EUR-1100 1.5 mg; EUR-1100 3.0 mg
Drug: placebo — matching placebo
  Arms: placebo

SUMMARY:
Eosinophilic esophagitis (EoE) is an inflammatory disease of the esophagus, characterized by eosinophilic infiltration and gastrointestinal (GI) symptoms. There are no pharmacological treatments for EoE approved by the US Food and Drug Administration (FDA). Supported by published case series and controlled trials in children and adults, the most widely used drug treatment for EoE is off-label use of corticosteroids intended for local (esophageal mucosal) action.

This study will evaluate the safety and tolerability of orally administered EUR-1100 once or twice daily. Eligible subjects will be randomized into one of the 3 treatment groups. The Treatment Period will be 8 weeks during which subjects will visit the clinic at the screening visit, randomization, week 4, 8 and 1 week after end of treatment for clinical symptom assessment and safety evaluation. Additional phone visits will occur at week 2 and week 6.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female subjects aged ≥ 12 and ≤ 55 years;
* Written informed consent (parent or guardian must sign when applicable) and assent form, if required;
* Evidence of eosinophilic esophagitis defined by esophageal mucosal eosinophil count greater than or equal to 24 per HPF (400x magnification) in at least 1 of the esophageal sites biopsied (proximal/middle and/or distal);
* Lack of histological response to previously administered high dose proton pump inhibitor;
* Clinical symptoms of eosinophilic esophagitis with at least one of the following symptoms: chest pain or discomfort, dysphagia (difficulty swallowing) or food impaction.

Key Exclusion Criteria:

* Known contraindication, hypersensitivity or intolerance to corticosteroids;
* Any physical, mental, or social condition, history of illness or laboratory abnormality that, in the investigator's judgment, might interfere with study procedures or the ability of the subject to adhere to and complete the study;
* Oral or esophageal mucosal infection of any type;
* Any condition affecting the esophageal mucosa or altering esophageal motility other than EoE;
* Use of systemic (oral or parenteral) or inhaled, intranasal or high-potency dermal topical corticosteroids in the 30 days prior to the esophageal biopsy required for entrance to this study (or prior to EGD if done during the pre-Screening period) or at any time between the biopsy and the Randomization Visit;
* Adrenal suppression;
* Any medical condition in which the use of anti-inflammatory or immunosuppressant drugs are required or may be anticipated to be required during the study;
* Contraindication to EGD or esophageal biopsy or narrowing of the esophagus precluding EGD;
* History of esophageal or gastric surgery (history of esophageal dilatation is allowed);
* Gastrointestinal bleeding;
* Current chronic infection, immunosuppression, immunodeficiency;
* History or presence of Crohn's disease, celiac disease, or other inflammatory disease of the gastrointestinal tract;
* Alcohol or drug abuse;
* Female subjects who are pregnant or breastfeeding;
* Participation in a clinical study involving an investigational drug within 30 days of the Screening Visit.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Morning serum cortisol (change from baseline measure) | Screening visit (up to 21 days), week 4, week 8 and follow-up
Standard safety laboratory tests | Screening visit (up to 21 days), week 4, week 8 and follow-up
  Hematology, serum chemistry and liver function tests, urinalysis, urine chemistry
Treatment-emergent adverse events collection | Screening visit (up to 21 days), Randomization day, week 2 and week 6(phone visit), week 4 and week 8 (office visit), follow-up (office visit, up to 11 days after week 8 visit)
Physical examination and vital signs collection | Screening (up to 21 days), week4, week 8 and follow-up

SECONDARY OUTCOMES:
Esophagoduodenoscopy with multiple biopsies | Screening (up to 21 days) and week 8
Patient reported outcomes, and physician global assessment | Screening (up to 21 days), week 4 and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Ikuo Hirano, MD, Principal Investigator — Northwestern University School of Medicine
Locations (7):
- United States (7):
  - Children's Center for Digestive Health, Atlanta, Georgia
  - Northwestern University School of Medicine, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - South Jersey Pediatric Gastroenterology, Mays Landing, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - O&O Alpan LLC Center for Clinical Trials, Fairfax, Virginia

REFERENCES:
- [Derived] Schoepfer AM, Hirano I, Coslovsky M, Roumet MC, Zwahlen M, Kuehni CE, Hafner D, Alexander JA, Dellon ES, Gonsalves N, Leung J, Bussmann C, Collins MH, Newbury RO, Smyrk TC, Woosley JT, Yang GY, Romero Y, Katzka DA, Furuta GT, Gupta SK, Aceves SS, Chehade M, Spergel JM, Falk GW, Meltzer BA, Comer GM, Straumann A, Safroneeva E; International EEsAI Study Group. Variation in Endoscopic Activity Assessment and Endoscopy Score Validation in Adults With Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1477-1488.e10. doi: 10.1016/j.cgh.2018.11.032. Epub 2018 Nov 23. PMID 30476587